CLINICAL TRIAL: NCT04296383
Title: A Randomized, Double-blind, Parallel-controlled,Multicenter Clinical Study of Xiyanping Injection Combined With Azithromycin and Azithromycin for Children With Pneumonia
Brief Title: Xiyanping Injection Combined With Azithromycin VS Azithromycin for Children With pneumoniaProtozoal Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QF-XYP1908-1
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Mycoplasma Pneumoniae Pneumonia
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin plus Xiyanping injection group (Experimental)
  Interventions: Drug: Azithromycin plus Xiyanping injection
- Azithromycin group (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin plus Xiyanping injection — Azithromycin for injection is 10mg / (kg • d), the maximum dose does not exceed 0.5g / d;Xiyanping injection intravenously, 0.4mL / (kg.d) daily, Qd
  Arms: Azithromycin plus Xiyanping injection group
Drug: Azithromycin — Azithromycin for injection is 10mg / (kg • d), the maximum dose does not exceed 0.5g / d
  Arms: Azithromycin group

SUMMARY:
Mycoplasma pneumoniae pneumonia in children is one of the major diseases in children's respiratory department in China, but there are still large clinical unmet needs.

DETAILED DESCRIPTION:
In order to further verify the clinical value and safety of Xiyanping injection in children with Mycoplasma pneumoniae pneumonia, to provide references for subsequent confirmatory research, and to provide more reasonable and standardized application guidance and basis for clinical practice, we intend to adopt more rigorous Scientific design to carry out a multi-center, randomized, double-blind, parallel-controlled study of Xiyanping injection in the treatment of children with Mycoplasma pneumoniae pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. 5 to 14 years of age at the time of screening;
2. Children who meet the Western medicine clinical diagnosis standard of Mycoplasma pneumoniae and the mycoplasma pneumoniae IgM antibody titer ≥1 : 80, or Mycoplasma pneumoniae DNA or RNA (PCR) test positive, or rapid identification of Mycoplasma pneumoniae antibodies positive;
3. Heat course ≤ 5 days;
4. The total number of peripheral blood routine leukocytes is within the normal range;
5. The child's legal guardian or / and himself voluntarily participate in the study, and the legal guardian agrees and signs the informed consent form (while children ≥8 years of age need to voluntarily sign the informed consent form);
6. According to the researcher's judgment, the subject / legal guardian is believed to be reliable and able to comply with this plan, visit plan and medication arrangement.

Exclusion Criteria:

1. Have a disease that needs to be distinguished from Mycoplasma pneumoniae pneumonia (MPP);
2. Patients with basic diseases such as primary immunodeficiency disease, acquired immunodeficiency syndrome, congenital respiratory malformation, abnormal lung development, aspiration pneumonia, lung malignancies, etc .;
3. Congenital abnormalities of heart and lung, combined with serious primary diseases such as cardiovascular, cerebrovascular, liver, kidney, and hematopoietic system, or any laboratory test indicators meet the following criteria: alanine aminotransferase (ALT), aspart Amino acid aminotransferase (AST)> 2.0 times, serum creatinine (Cr)> 1.5 times the upper limit of normal value (ULN);
4. Those who have been diagnosed with Mycoplasma pneumoniae in the past 3 months;

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2021-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Clinical recovery time | up to day 19
  Time from study drug use to complete fever and cough relief, measured in days